CLINICAL TRIAL: NCT01124383
Title: The Impact of Anesthesia on the Absorption of Glycine in Operative Hysteroscopy: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Association of Professors of Obstetrics and Gynaecology of Canada (Other)
Responsible Party: Marie-Eve Bergeron MD, Centre Hospitalier Universitaire de Québec, Université Laval
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUQ: 118.05.07; CHA: CER-019-001 (Other: Centre Hospitalier Universitaire Affilié de Québec)
Record Dates: First submitted 2010-04-13; First posted 2010-05-17 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-04

CONDITIONS: The Absorption of Glycine in Operative Hysteroscopy
Keywords: Glycine absorption; Operative hysteroscopy; Endometrial resection; General anesthesia; Local anesthesia
MeSH Terms: interventions — Anesthesia, General; Midazolam; Sufentanil; Propofol; Rocuronium; Sevoflurane; Ephedrine; Anesthesia, Local; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General anesthesia (Active Comparator)
  Interventions: Procedure: General anesthesia
- Local anesthesia with sedation (Active Comparator)
  Interventions: Procedure: Local anesthesia with sedation

INTERVENTIONS:
Procedure: General anesthesia — For women in the general anesthesia group, general anesthesia is induced using midazolam 1-3 mg, sufentanil 0.15-0.25 mcg/kg and propofol 1-3 mg/kg. Rocuronium 0.6 mg/kg is allowed. Anesthesia is maintained with sevoflurane titrated to maintain a blood pressure within 20% of preoperative normal and, if needed, ephedrine can be used for this purpose. Patients are ventilated in a normocapnic range with a positive end-expiratory pressure of 3 to 5 mmHg.
  Other Names: Midazolam; Sufentanil; Propofol; Rocuronium; Sevoflurane; Ephedrine
  Arms: General anesthesia
Procedure: Local anesthesia with sedation — For women in the local anesthesia group a paracervical block is performed by the gynecologist using a total of 20 mL of 1% lidocaine intracervically at 2, 4, 7 and 10 o'clock positions and in the area of uterosacral ligaments. Once the block completed, the surgeon waits at least five minutes before performing cervical dilatation to allow for sufficient analgesia. Intravenous sedation consists of midazolam, sufentanil and propofol administered by the anesthesiologist in sufficient doses to maintain a spontaneous ventilation with a Ramsay score < 4.
  Other Names: Lidocaine; Midazolam; Sufentanil; Propofol
  Arms: Local anesthesia with sedation

SUMMARY:
This study aimed to compare two types of anesthesia (general anesthesia and local anesthesia with sedation) on the absorption of glycine in operative hysteroscopy.

DETAILED DESCRIPTION:
As a minimally invasive procedure, operative hysteroscopy has gained popularity in the past two decades and became a standard surgical treatment for abnormal uterine bleeding unresponsive to medical management. Despite its increasing use, little information is known on the predictors of its potential complications. The absorption of glycine has been reported as the most common complication of this procedure and it remains an unpredictable complication that may lead to life-threatening conditions.

This randomized controlled trial is conducted in two centers: a tertiary care center and in a community hospital over a period of 18 months. This study aimed to compare two types of anesthesia on the absorption of glycine in operative hysteroscopy. Eligible patients undergoing operative hysteroscopy for abnormal uterine bleeding are randomized in two groups: group general anesthesia and group local anesthesia with sedation.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal uterine bleeding with clinical indication for operative hysteroscopy according to an obstetrician-gynecologist.
* American Society of Anesthesia (ASA) class 1 or 2

Exclusion Criteria:

* Any contraindications to hysteroscopy (suspicion of pelvic or vaginal-cervical infection, severe hemorrhage, pregnancy, suspicion of neoplasia and previous uterine perforation)
* ASA class 3 or more
* Women who had a previous endometrial resection
* Diabetic patients
* Women requiring a predetermined type of anesthesia because of a specific medical condition

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Median absorption of glycine (10th-90th centile) | The absorption of glycine is measured between time of the introduction of the resectoscope and its final withdrawal. Assessed between 1 minute and 20 minutes after the end of surgery
  The primary outcome is the median absorption of glycine (10th-90th centile). The glycine absorption is measured by an automated surgical irrigator (tandem canister: Equimat and Endomat; Karl Storz Endoscopy, Tuttlingen, Germany) and it represent the difference between the input and the output of glycine used for the irrigation of the uterine cavity.

SECONDARY OUTCOMES:
Absorption of glycine greater than 1000 mL | The absorption of glycine is measured between time of the introduction of the resectoscope and its final withdrawal. Assessed between 1 minute and 20 minutes after the end of surgery
  The total absorption of glycine is measured by an automated surgical irrigator (tandem canister: Equimat and Endomat; Karl Storz Endoscopy, Tuttlingen, Germany).
Discontinuation of surgery because of excessive absorption. | Assessed between 1 minute and 20 minutes after the end of surgery
  Left at the discretion of the surgeon and anesthesiologist. However, according to the guidelines of the ACOG and the AAGL, it is recommended to stop the surgery when the glycine deficit exceeds 1000-1500 mL. Therefore, the surgeon who is blinded to the absorption rate will be informed when it reachs 500 and 1000 mL.
Difference of natremia pre and post-procedure | Assessed the same day of surgery (no more than 6 hours after surgery)
  In the hour preceeding the surgery and in the hour following surgery, natremia will be measured in the patient serum.
Postoperative severe hyponatremia | Assessed the same day of surgery (no more than 6 hours after surgery)
  Defined as a patient's natremia below 125 meq/L in the first postoperative hour.
Patient's satisfaction towards the type of anesthesia | Assessed on postoperative day one. In average 24 hours after surgery.
  Patient's satisfaction toward their anesthesia was evaluated by the following yes or no question: "If you had to undergo the same surgery, would you choose the same type of anesthesia?".
Quality of life and recovery | Assessed on postoperative day one. In average 24 hours after surgery.
  8-item Short-Form Health Survey (SF-8) standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bujold, MD MSc FRCSC, Study Chair — Centre hospitalier universitaire de Québec- Université Laval; Marie-Eve Bergeron, MD, Principal Investigator — Centre hospitalier universitaire de Québec- Université Laval; Pascale Ouellet, MD, Principal Investigator — Centre hospitalier universitaire de Québec- Université Laval
Locations (1):
- Centre Hospitalier Universitaire de Québec, Québec, Quebec, Canada